CLINICAL TRIAL: NCT05747521
Title: A Single Arm, Single Center, Prospective Clinical Study of Anrotinib Hydrochloride Combined With Doxorubicin in the Neoadjuvant Treatment of High-grade Soft Tissue Sarcoma
Brief Title: Anrotinib Hydrochloride Combined With Adriamycin for Neoadjuvant Treatment of High-grade Soft Tissue Sarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, YaoWeitao, Chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-STS-001
Record Dates: First submitted 2023-02-14; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anrotinib hydrochloride combined with adriamycin (Experimental): Anrotinib hydrochloride combined with adriamycin neoadjuvant therapy for patients with high-grade soft tissue sarcoma
  Interventions: Drug: Anrotinib hydrochloride combined with adriamycin

INTERVENTIONS:
Drug: Anrotinib hydrochloride combined with adriamycin — To evaluate the efficacy of anrotinib hydrochloride combined with doxorubicin in the neoadjuvant treatment of high-grade soft tissue sarcoma

SUMMARY:
This is an investigator-initiated, single-arm, single-center, prospective clinical study with an estimated 58 patients enrolled to explore the efficacy and safety of anrotinib hydrochloride in combination with doxorubicin and radiotherapy in patients with high-grade soft tissue sarcoma.

DETAILED DESCRIPTION:
This is a single-arm, single-center, prospective investigator-initiated clinical study of 58 patients enrolled in Henan Cancer Hospital to explore the efficacy and safety of anrotinib hydrochloride combined with doxorubicin and radiotherapy in patients with high-grade soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old, regardless of gender.
2. Patients with soft tissue sarcomas of trunk or limbs of G3 confirmed by histology or cytology; Pathological types include synovial sarcoma, undifferentiated pleomorphic sarcoma, leiomyosarcoma and fibrosarcoma.
3. No treatment with anthracyclines or anti-angiogenic targeted drugs.
4. According to RECIST Version 1.1 (Annex 1), there were measurable lesions at baseline with primary tumors larger than 5cm and poor location in deep fascia;
5. ECOG Physical status score (Annex 2) a is 0-2, and the expected survival period is more than 6 months.
6. Recovery from previous treatment: According to NCI-CTCAE version 5.0, all side effects (except hair loss) resolved to grade 1 or below.
7. If the major organs are functioning normally, the following criteria are met:

   Hemoglobin (Hb) ≥ 95g/L, Neutrophil (ANC) ≥1.5×109/L, Platelet count (PLT) ≥ 80×109/L, Serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN), blood urea nitrogen (BUN) ≤ 2.5× upper limit of normal (ULN); Total bilirubin (TB) ≤ 1.5ULN; Aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; Albumin (ALB) ≥ 35 g/L Prothrombin time (PT) and partial prothrombin time (PTT) ≤1.2×ULN Left ventricular ejection fraction ≥50% Blood pressure was controlled within 140/90 mmHg before enrollment
8. Women of childbearing age must have been using reliable contraception or have had a pregnancy test (serum or urine) with negative results within 7 days prior to inclusion and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last test drug administration. For men, consent is required to use an appropriate method of contraception or to have been surgically sterilized during the trial period and within 8 weeks after the last administration of the trial drug
9. Sign an informed consent form (or legal representative sign) to demonstrate that they understand the purpose of the study and the procedures required by the Institute, and are willing to participate in the study.

Exclusion Criteria:

1. Previous exposure to antirotinib hydrochloride or other small molecule anti-angiogenic TKI drugs, or anti-angiogenic mab drugs (such as Sunitinib, Sorafenib, bevacizumab, imatinib, Famitinib, Apatinib, Regafenib, etc.).
2. Systemic antitumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks prior to treatment with the experimental drug) was planned for 4 weeks prior to enrollment or during the medication period of this study. Over extended field radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment.
3. Other malignant neoplasms (other than squamous cell carcinoma of skin) in the past 3 years;
4. Imaging (CT or MRI) showed that the tumor lesions had tumors invading local great vessels, or were accompanied by tumor thrombus formation of large veins (iliac vessels, inferior vena cava, pulmonary veins, superior vena cava);
5. Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral therapy;
6. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal medical treatment);
7. Urine routine indicated urine protein ≥ ++, or confirmed 24 hours urine protein volume ≥1.0 g, urine protein/creatinine ≥1;
8. Uncontrolled co-morbidity, including, but not limited to, poorly controlled diabetes, persistent active infections, or mental illness or social conditions that may affect study compliance;
9. Abnormal coagulation function (INR > 1.5 or PT >1.2 ULN or PTT >1.2 ULN), bleeding tendency or receiving thrombolytic or anticoagulant therapy; Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their equivalents;
10. Obvious blood coughing or daily hemoptysis of 2.5ml or above within 2 months before enrollment;
11. Subjects with any medical conditions that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, such as active gastrointestinal ulcers, known luminal metastases, inflammatory bowel disease, and a history of abdominal fistula, gastrointestinal perforation, or abdominal abscess within 28 days prior to study initiation;
12. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction, including but not limited to a history of stomach or small intestine resection, and malabsorption syndrome;
13. Subjects who have had any of the following cardiovascular diseases in the past six months: Stroke (CVA) or transient cerebral ischemia (TIA), arrhythmia (including QTc interval ≥450 ms for men and 470 ms for women), angina, coronary angiogenesis or heart stents, pulmonary embolism, Patients with untreated or anticoagulant therapy for less than 6 weeks with deep vein thrombosis, arterial thrombosis, Grade III or IV heart failure as defined by the New York Heart Association's functional grading system, and clinically significant pericardial disease in patients with left ventricular ejection fraction (LVEF) < 50% indicated by cardiac color ultrasound, Or electrocardiogram suggests acute ischemia or abnormal conduction system;
14. Patients with active viral hepatitis B or hepatitis C, or active infections requiring antimicrobial treatment (e.g. antibiotics, antiviral drugs, antifungal drugs); 15.4 weeks of participation in other antitumor clinical trials (non-immunotherapeutic;

16. Hypothyroidism patients: TSH>4.2mlU/L; 17.7 days of treatment with a potent CYP3A4 inhibitor, or 12 days prior to study entry. Drugs with substrates for CYP3A4, CYP2D6, or CYP2C8 should be avoided; 18.4 weeks use of drugs that may lead to prolonged QT interval and tip torsion; 19. Open wounds, sores or fractures; 20.4 weeks of surgery; 21. Serous effusion (including pleural effusion, ascites, pericardial effusion) with clinical symptoms that require surgical treatment; 22. Known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulation disorders, thrombocytopenia, hyperplenism, etc.); 23. Lactation period; 24. Hiv-positive patients; 25. Those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders; 26. Any condition that the investigator considers to be prejudicial to the subject or to the subject's inability to meet or perform the study requirements exists.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | It is expected to take up to 60 months from treatment to disease progression
  Proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No